CLINICAL TRIAL: NCT02997345
Title: Patient Registry for Women Diagnosed With Preterm Premature Rupture of Membranes or PPROM During Pregnancy
Brief Title: PPROM Registry (Preterm Premature Rupture of Membranes)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American Alliance for pProm Support (Other)
Responsible Party: Principal Investigator, Erin Thatcher, Director, American Alliance for pProm Support
Other Study IDs: tpr072013
Record Dates: First submitted 2016-10-18; First posted 2016-12-20 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes; Oligohydramnios; Premature Birth
Keywords: PPROM
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes; Oligohydramnios; Premature Birth

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PPROM (Preterm Premature Rupture of Membranes): PPROM / Preterm Premature Rupture of Membranes <37 weeks
  Interventions: Other: There is no intervention associated with this study.

INTERVENTIONS:
Other: There is no intervention associated with this study. — There is no intervention associated with this study.

SUMMARY:
Preterm Premature Rupture of Membranes (PPROM) before 37 weeks of pregnancy is responsible for 40% of preterm births in the United States. The PPROM Registry aims to identify possible causes of PPROM, evaluate trends in expectant management, measure maternal and fetal care, and to review short term and long term outcomes of affected pregnancies and births.

DETAILED DESCRIPTION:
Detailed Description

Preterm Premature Rupture of Membranes (pProm) is a factor in 40% of preterm births. The earlier in pregnancy pProm occurs, the greater the potential latency period. Threats to the pregnancy include placental abruption, umbilical cord prolapse, infection, and insufficient pulmonary development, and preterm delivery. Management of pProm may include immediate delivery, induction, or expectant management.

It is still unclear what is considered best practice for the course of treatment in pProm pregnancies and post- delivery care of pProm babies in Neonatal Intensive Care Units (NICU), as well as the long term outcomes of pProm survivors. Unfortunately, there are few recent studies available for review and those that exist often do not reflect the current treatments or innovations that have taken place, especially in neonatal care. Many of the studies available focusing on pProm have very small sample sizes, as well as very short follow-up post-delivery, resulting in a wide range of reported outcomes, especially regarding the morbidity and mortality associated with pProm.

The pProm registry is the first of its kind and will provide a large cohort of data for study. The purpose of this registry is to better understand pregnancies and births impacted by pProm. This includes how pProm is managed in pregnancy and in how pProm neonates are cared for in the NICU; identifying trends in expectant management, and to detect short term and long term outcomes of those affected.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Preterm Premature Rupture of Membranes (PPROM) prior to 37 weeks of pregnancy

Exclusion Criteria:

* Those without a clinical diagnosis or confirmation of PPROM in pregnancy
* Diagnosis of PROM beyond 37 weeks of pregnancy

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women diagnosed with Preterm Premature Rupture of Membranes (PPROM) prior to 37 weeks of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Early Neonatal Mortality Rate | 28 days post delivery

SECONDARY OUTCOMES:
Stillbirth / Perinatal Mortality Rate | Upon delivery

OTHER OUTCOMES:
Review of Socio-Economic Factors in pProm | Single assessment (observational) at conclusion of pregnancy +30 days, monitored for up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- Www.Aapprom.Org/the-Registry, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: PPROM Registry — https://www.aapprom.org/the-registry